CLINICAL TRIAL: NCT02774278
Title: MERIT - A Phase II Marker Identification Trial for Tarceva in Second Line NSCLC Patients
Brief Title: A Study of Erlotinib (Tarceva) in Participants With Non-Small Cell Lung Cancer (NSCLC)
Acronym: MERIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO18279; 2004-005096-42 (EudraCT Number)
Record Dates: First submitted 2016-05-03; First posted 2016-05-17 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- Erlotinib (Experimental): Participants will receive erlotinib orally daily until disease progression, unacceptable toxicity or death.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib will be administered at 150 milligrams (mg) orally daily until disease progression, unacceptable toxicity or death.
  Other Names: Tarceva

SUMMARY:
This study will assess potentially predictive markers of efficacy in participants with NSCLC receiving oral erlotinib (Tarceva) therapy. The anticipated time on study treatment is until disease progression, unacceptable toxicity or death.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC
* Tumor accessible for biopsy by bronchoscopy
* Disease progression following course of standard chemotherapy, or participants unwilling/unable to undergo chemotherapy

Exclusion Criteria:

* Unstable systemic disease
* Any other malignancies in the last 5 years
* Brain metastases
* Previous treatment with therapy acting on the epidermal growth factor receptor (EGFR) axis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2005-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (22):
- Brussels, Belgium
- Sofia, Bulgaria
- Estonia (2):
  - Tallinn
  - Tartu
- France (2):
  - Montpellier
  - Paris
- Germany (2):
  - Cologne
  - Großhansdorf
- Hong Kong, Hong Kong
- Dublin, Ireland
- Perugia, Italy
- Poland (4):
  - Gdansk
  - Lodz
  - Lublin
  - Poznan
- Russia (2):
  - Moscow
  - Saint Petersburg
- Singapore, Singapore
- Spain (2):
  - Barcelona
  - Madrid
- Taipei, Taiwan
- Weston-super-Mare, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib: Erlotinib was administered at 150 milligrams (mg) orally daily until disease progression, unacceptable toxicity or death.
Period: Overall Study
Arm/Group | Erlotinib
Started | 264
Safety Analysis Population (SAP) | 261 (SAP: all participants who received at least 1 dose of trial medication and had a safety follow-up.)
Completed | 0
Not Completed | 264
Not completed — Lack of Efficacy | 199
Not completed — Death | 29
Not completed — Adverse event/intercurrent illness | 16
Not completed — Refused treatment/did not cooperate | 9
Not completed — Administrative reasons | 6
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants.
Arm/Group | Erlotinib
Number analyzed (Participants) | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 184

OUTCOME MEASURES:

1. Primary Outcome: Number of Differentially Expressed Genes Associated With Clinical Benefit
Description: Affymetrix gene expression profiles were primarily analyzed to identify differentially expressed genes between the participants who derived clinical benefit status and those who did not. Analysis was performed using a multivariate linear model (with clinical benefit status, histology, ethnicity, sex, RNA integrity number (RIN), smoking status and stage as predictors), and a False Discovery Rate criteria of below 0.3 as cut-off. Clinical benefit is defined in the Outcome Measure 5.
Time Frame: Baseline until disease progression, unacceptable toxicity or death, evaluated up to 4 years
Population: Primary analysis set (PAS) included all participants who provided evaluable tissue samples and were included in the primary Affymetrix efficacy analysis.
Measure: Number; unit: genes
Arm/Group | Erlotinib
Number analyzed (Participants) | 102
genes | 0

2. Primary Outcome: Number of Epidermal Growth Factor Receptor (EGFR) Mutation Participants Who Achieved Clinical Benefit
Description: Affymetrix gene expression profiles were primarily analyzed to identify differentially expressed genes between the participants who derived clinical benefit status and those who did not. Analysis was performed using a multivariate linear model (with clinical benefit status, histology, ethnicity, sex, RNA integrity number (RIN), smoking status and stage as predictors), and a False Discovery Rate criteria of below 0.3 as cut-off. Number of participants with EGFR mutation (L858R/ exon 19 deletion) and who achieved clinical benefit status was reported. Clinical benefit is defined in the Outcome Measure 5.
Time Frame: Baseline until disease progression, unacceptable toxicity or death, evaluated up to 4 years
Population: PAS participants who had EGFR mutation at baseline were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 6
participants | 6

3. Primary Outcome: Number of KRAS Mutation Participants Who Achieved Clinical Benefit
Description: Affymetrix gene expression profiles were primarily analyzed to identify differentially expressed genes between the participants who derived clinical benefit status and those who did not. Analysis was performed using a multivariate linear model (with clinical benefit status, histology, ethnicity, sex, RNA integrity number (RIN), smoking status and stage as predictors), and a False Discovery Rate criteria of below 0.3 as cut-off. Number of participants with KRAS gene mutation and who achieved clinical benefit status was reported. Clinical benefit is defined in the Outcome Measure 5.
Time Frame: Baseline until disease progression, unacceptable toxicity or death, evaluated up to 4 years
Population: PAS participants who had KRAS mutation at baseline were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 10
participants | 4

4. Secondary Outcome: Percentage of Participants With Overall Response of Complete Response (CR) or Partial Response (PR) Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Tumor response was defined as either a CR or a PR prior to failure (disease progression, death from any cause, or a second malignancy). CR was defined as the complete disappearance on magnetic response imaging of all enhancing tumor and mass effect on a stable or decreasing dose of dexamethasone (or only receiving adrenal replacement doses) accompanied by a stable or improving neurologic examination that was maintained for at least 12 weeks. PR was defined as a greater than or equal to 50 percent (%) reduction in tumor size by bi-dimensional measurement on a stable or decreasing dose of dexamethasone accompanied by a stable or improving neurologic examination that was maintained for at least 12 weeks.
Time Frame: Baseline until disease progression, unacceptable toxicity or death, evaluated up to 4 years
Population: Analysis population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 264
percentage of participants | 15.2 [11.1 to 20.1]

5. Secondary Outcome: Percentage of Participants With Clinical Benefit (CR, PR, or Stable Disease [SD] for at Least 12 Weeks After Study Entry) Using RECIST
Description: Clinical benefit was defined as either a CR, PR, or SD prior to failure (disease progression, death from any cause, or a second malignancy). CR: complete disappearance on magnetic response imaging of all enhancing tumor and mass effect on a stable or decreasing dose of dexamethasone (or only receiving adrenal replacement doses) accompanied by a stable or improving neurologic examination that was maintained for at least 12 weeks. PR: greater than or equal to 50% reduction in tumor size by bi-dimensional measurement on a stable or decreasing dose of dexamethasone accompanied by a stable or improving neurologic examination that was maintained for at least 12 weeks. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference smallest sum of longest dimensions since treatment started associated to non-progressive disease response for non-target lesions. PD: unequivocal progression of existing non-target lesions.
Time Frame: Baseline until disease progression, unacceptable toxicity or death, evaluated up to 4 years
Population: Analysis population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 264
percentage of participants | 31.4 [25.9 to 37.4]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Safety analysis population (SAP) included all participants who received at least one dose of the trial medication and had a safety follow-up.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 65/261
Other Adverse Events (participants affected / at risk) | 209/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=261)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Asthenia (General disorders) | 3
General physical health deterioration (General disorders) | 3
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1
Agitation (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Arterial haemorrhage (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=261)
Rash (Skin and subcutaneous tissue disorders) | 133
Dry skin (Skin and subcutaneous tissue disorders) | 33
Pruritus (Skin and subcutaneous tissue disorders) | 32
Acne (Skin and subcutaneous tissue disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 84
Vomiting (Gastrointestinal disorders) | 26
Nausea (Gastrointestinal disorders) | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 39
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 15
Fatigue (General disorders) | 32
Pyrexia (General disorders) | 14
Anorexia (Metabolism and nutrition disorders) | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.